CLINICAL TRIAL: NCT03195686
Title: Efficacy of PLEM100(Inbody®) to Measure the the Sedation Level in Pediatric Patients
Brief Title: Efficacy of PLEM100(Inbody®) in Children
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: 1795-110-855
Record Dates: First submitted 2017-06-18; First posted 2017-06-22 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Development, Child

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PLE100(Inbody®) — PLE100(Inbody®) monitoring in children to be operated under the total intravenous anesthesia (Propofol)

SUMMARY:
Evaluation of efficacy of PLEM100(Inbody®) in measuring the sedation level in pediatric patients

DETAILED DESCRIPTION:
The investigators plan to gather the basic data relevant to measurement of the level of consciousness/sedation in pediatric patients with developing brain by using PLEM100(Inbody®)

PLEM100 (Inbody®) is a medical equipment to measure, based on phase lag entropy algorithm, the level of patient consciousness, which is expressed by PLE score ranging from 0 (burst suppression or deep sedated) to 100 (awake).

In this study, pediatric patients aged from 3 to 6 years old who undergo total intravenous general anesthesia are chosen as target subjects. The investigators measure how PLE score changes during 1) anesthesia induction, 2) anesthesia maintenance, 3) emergence from anesthesia. Then, the PLE score would be validated by analyzing the correlation with the consciousness level expressed in University of Michigan Sedation Scale (UMSS).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients to be operated under general anesthesia, aged from 3 to 6 years
* Written Consent is available from a parent who has been explained about the study
* Elective surgery

Exclusion Criteria:

* Patients who cannot be attached by PLEM100 (Inbody®) sensors to the forehead or the side of the head
* Patients Having Cerebral Vascular Diseases in the past or present
* Patients with Developmental delay
* Patients to be admitted to intensive care unit or sedated after receiving operation
* Patients who researchers decide are not eligible to be enrolled in the study because of various factors including clinical test results.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients to be operated under general anesthesia, aged from 3 to 6 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
PLE100 score (0 to 100) | baseline and end of surgery
  Changes of PLE100 score

SECONDARY OUTCOMES:
The level of consciousness measured in University of Michigan Sedation Scale (UMSS) | baseline and end of surgery
  correlation with the PLE100 scores and concentraion of propofol
pharmacodynamic model | baseline and end of surgery
  UMSS with propofol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jang YE, Ji SH, Lee JH, Kim EH, Kim JT, Kim HS. The relationship between the effect-site concentration of propofol and sedation scale in children: a pharmacodynamic modeling study. BMC Anesthesiol. 2021 Sep 9;21(1):222. doi: 10.1186/s12871-021-01446-y. PMID 34503455